CLINICAL TRIAL: NCT01389388
Title: Cholesterol Plaques in Carotid and Coronary Arteries and the Effect of Rosuvastatin in Rheumatoid Arthritis, Ankylosing Spondylitis and Other Inflammatory Joint Diseases
Brief Title: Effects of Rosuvastatin on Carotid Artery Plaques in Patients With Inflammatory Joint Disease
Acronym: RORAAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Anne Grete Semb, Leader of the Preventive Cardio-Rheuma clinic, Diakonhjemmet Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2009/2219; 2008-005551-20 (EudraCT Number)
Record Dates: First submitted 2010-04-16; First posted 2011-07-08 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Carotid Artery Plaque; Ankylosing Spondylitis; Rheumatoid Arthritis
Keywords: Carotid plaques; inflammatory joint disease; statins; inflammation; lipoprotein components
MeSH Terms: conditions — Carotid Stenosis; Spondylitis, Ankylosing; Arthritis, Rheumatoid; Inflammation | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin intervention (Experimental): Patients > 70 years will be given Rosuvastatin of 5 mg a day, uptitering the dose until the LDL level of 1.6-1.8 mmol/l has been reached. Patient <70 years, strat on Rosuvastatin 20 mg a day, uptitered to 40 mg a day, with the LDL of 1.6-1.8 mmol/l. -1.8 mmol/l. The objective is that all the participants should have reached a LDL level of 1.6-1.8 mmol/l 3 months after the start of the study. The participants will remain on Rosuvastatin medication for a total of 18 months.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — All the patients who have signed the informed consent will after they have had performed a MCT and possibly SCC with an IVUS, will be give Rosuvastatinuntill their LDL level has reached 1.6-1.8 mmol/l. The objective is that all the participants should have reached 1.6-1.8 mmol/l 3 months after the start of the study. The participants will remain on Rosuvastatin medication for a total of 18 months.
  Other Names: Brand name for Rosuvastatin is Crestor

SUMMARY:
Patients with rheumatoid Arthritis (RA) and Ankylosing Spondylitis (AS) are at greater risk of developing cardiovascular disease. The reason(s) for this have not been well investigated, but there is a general understanding that systemic inflammation plays a part in the increased cardiovascular morbidity and mortality. In spite of the increased risk in these patients, they have not been included as a high risk patient group in cardiovascular prevention guidelines.

The investigators have carried out a cardiovascular study of RA and AS patients, as well as patients with arthritis for the first time. The investigators have demonstrated cholesterol plaques in the carotid artery in some of these patients. Plaques in the carotid artery represent a risk for development of cerebral stroke and are significantly associated with myocardial infarction. These plaques, which are asymptomatic and do not cause haemodynamically significant narrowing, diameter reduction (i.e. operation is not indicated), are vascular atheromatous disease. Therefore, according to prevailing cardiovascular guidelines (SCORE 2007), these patients shall have secondary prevention with a lipid lowering agent with the LDL-cholesterol goal of 1.8 mmol/L and HDL-cholesterol > 1.0 mmol/L for men and > 1.1 mmol/L for women.

Statins are cholesterol-lowering drugs, and have been shown to reduce the risk of cardiovascular disease significantly. In addition, reduction in the size of coronary plaques has been induced by statins, when the LDL has been reduced to 1.6-1.8 mmol/l. Plaques in the carotid or coronary arteries have not previously been treated and characterized in patients with RA, AS and other inflammatory forms of arthritis.

The aim of this study is to treat patients with cholesterol plaques in the carotid artery with cholesterol-lowering medication, in the form of Rosuvastatin for 18 months, and characterize the effects on the plaques in the carotid and coronary arteries. In addition, the investigators want to clarify the connection between plaques in the carotid and coronary arteries in patients with RA, AS and other inflammatory forms of arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men with RA, AS and other inflammatory forms of arthritis, aged 35-80 years.
2. Cholesterol plaques demonstrated in carotid artery by ultrasound.
3. Informed consent.

Exclusion Criteria:

1. Concomitant statin treatment
2. Arterial fibrillation or others with chronic irregular heart rhythm (because of CT).
3. Contraindication to statin treatment.

   * Hypersensitivity to statins
   * Liver disease with ASAT/ALAT ≥ twice the upper normal limit
   * Previous statin-induced myopathy or severe hypersensitivity reactions to other statins
   * Raised creatinine (because of contrast medium)
   * Pregnancy or breast feeding
   * Fertile women who do not use contraceptives
   * Cyclosporine treatment
   * Treatment with medicinal products that have a known interaction with Rosuvastatin
   * Uncontrolled hypothyroidism defined as TSH > 1.5 times ULN at the first visit (because of the connection between myopathy and hypothyroidism with statin treatment)
   * Creatinine clearance < 30 ml/min and <60 ml/min with a Rosuvastatin dose of 40 mg per day
4. Secondary hyperlipidemia

   * Primary hyperthyroidism
   * Nephrotic syndrome, creatinine > 2 mg/dl
   * Uncontrolled diabetes mellitus (HbA1C > 10 %)
   * Plasma Triglycerides > 6.8 mmol/l
5. Other diseases or treatment that reduces the safety, or treatment with Rosuvastatin which would interfere with the end points of the study

   * Heart failure: NYHA class III B/IV
   * Haemodynamically significant valve defects
   * Established statin treatment
   * Gastrointestinal disease/treatment that can give malabsorption of Rosuvastatin
   * Cancer
   * Severe psychiatric disease
   * Life-threatening ventricular arrhythmias
   * Other medication that increases the risk of rhabdomyolysis
   * Known abuse of alcohol
   * Participation in other studies

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Carotid artery cholesterol plaque regression and stabilization | 18 months
  Reduction of plaque area and change of the plaque morphology to less vulnerable for rupture after 18 months with 40 mg Rosuvastatin daily.

SECONDARY OUTCOMES:
Disease activity and health measures, lipoprotein components and inflammatory biomarkers | 18 months
  Disease activity and Health status i. Disease activity will be measured by: 28-swollen-joint count, AIMS2, BASDAI ii. Health status will be measured by MHAQ, BASFI, Pain VAS, Fatigue VAS, life quality (HRQoL)
Carotid artery cholesterol plaque regression and stabilization | 18 months
  Lipoprotein components: Lipids, apolipoproteins, magnitude and functional measurements of these, for example of HDL
Carotid artery cholesterol plaque regression and stabilization | 18 months
  Biomarkers/inflammation parameters

CONTACTS AND LOCATIONS:
Overall Officials: Anne G Semb, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Anne Grete Semb, Department of Rheumatology, Diakonhjemmet hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Os HA, Rollefstad S, Gerdts E, Kringeland E, Ikdahl E, Semb AG, Midtbo H. Preclinical cardiac organ damage during statin treatment in patients with inflammatory joint diseases: the RORA-AS statin intervention study. Rheumatology (Oxford). 2020 Dec 1;59(12):3700-3708. doi: 10.1093/rheumatology/keaa190. PMID 32386421
- [Derived] Svanteson M, Rollefstad S, Klow NE, Hisdal J, Ikdahl E, Semb AG, Haig Y. Associations between coronary and carotid artery atherosclerosis in patients with inflammatory joint diseases. RMD Open. 2017 Sep 17;3(2):e000544. doi: 10.1136/rmdopen-2017-000544. eCollection 2017. PMID 28955501
- [Derived] Ikdahl E, Rollefstad S, Hisdal J, Olsen IC, Pedersen TR, Kvien TK, Semb AG. Sustained Improvement of Arterial Stiffness and Blood Pressure after Long-Term Rosuvastatin Treatment in Patients with Inflammatory Joint Diseases: Results from the RORA-AS Study. PLoS One. 2016 Apr 19;11(4):e0153440. doi: 10.1371/journal.pone.0153440. eCollection 2016. PMID 27093159
- [Derived] Ikdahl E, Hisdal J, Rollefstad S, Olsen IC, Kvien TK, Pedersen TR, Semb AG. Rosuvastatin improves endothelial function in patients with inflammatory joint diseases, longitudinal associations with atherosclerosis and arteriosclerosis: results from the RORA-AS statin intervention study. Arthritis Res Ther. 2015 Oct 8;17:279. doi: 10.1186/s13075-015-0795-y. PMID 26445924
- [Derived] Rollefstad S, Ikdahl E, Hisdal J, Olsen IC, Holme I, Hammer HB, Smerud KT, Kitas GD, Pedersen TR, Kvien TK, Semb AG. Rosuvastatin-Induced Carotid Plaque Regression in Patients With Inflammatory Joint Diseases: The Rosuvastatin in Rheumatoid Arthritis, Ankylosing Spondylitis and Other Inflammatory Joint Diseases Study. Arthritis Rheumatol. 2015 Jul;67(7):1718-28. doi: 10.1002/art.39114. PMID 25778850